CLINICAL TRIAL: NCT02607722
Title: The Special Drug Use-results Survey (All-Case Surveillance) of Ofev® Capsules in Patients With Idiopathic Pulmonary Fibrosis (IPF) in Japan
Brief Title: All-Case Surveillance of Ofev in Patients With IPF in Japan
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199.202
Record Dates: First submitted 2015-09-02; First posted 2015-11-18 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- IPF patients receiving Nintedanib: Patients diagnosed with idiopathic pulmonary fibrosis (IPF) based upon the most recent ATS/ERS/JRS/ALAT guideline and who initiated treatment with Ofev Capsules after the launch were registered into this study basically within 14 days from initiation of Ofev Capsules (from October 2015 to May 2023).
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib

SUMMARY:
This is a non-interventional study based on new data collection to gather real-world information (i.e., data under routine medical practice) on safety and effectiveness of the Ofev® Capsules treatment.

The study will consist of a baseline visit and follow-up visits at Week 4, 13, 26, 39, 52, 65, 78, 91 and 104 for patients who have newly initiated Ofev® Capsules. The patients will be followed up until discontinuation of Ofev® Capsules treatment.

As this is an observational study, no specific treatment is mandated or withheld from the patients. The choice of maintenance treatment for IPF must be according to regular medical practice and at the discretion of the physician (i.e., no randomised assignment of patient to treatment is performed).

All patients administrated Ofev® Capsules after the launch at the sites contracted with the sponsor will be registered. The Case Report Forms (CRFs) of 1000 patients will be collected. However the patient registration continues until the approval condition has been removed.

Patients participating in the subsequent follow-up will undergo regular observations. These observations should be reported after approximately Week 4, 13, 26, 39, 52, 65, 78, 91 and 104 since the initiation of Ofev® Capsules as long as they continue to receive the treatment. Patients will not be followed any longer once they are reported to have discontinued the Ofev® Capsules treatment.

ELIGIBILITY:
Inclusion criteria:

Essentially, patients are diagnosed with IPF based upon the most recent the American Thoracic Society (ATS), the European Respiratory Society (ERS), the Japanese Respiratory Society (JRS), and the Latin American Thoracic Association (ALAT) guideline.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1000 Japanese patients with IPF
Sampling Method: Non-Probability Sample
Enrollment: 10117 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Inoue Y, Ogura T, Azuma A, Kondoh Y, Homma S, Muraishi K, Ikeda R, Ochiai K, Sugiyama Y, Nukiwa T. Real-World Safety, Tolerability and Effectiveness of Nintedanib in Patients with Idiopathic Pulmonary Fibrosis: Final Report of Post-marketing Surveillance in Japan. Adv Ther. 2025 Feb;42(2):1075-1093. doi: 10.1007/s12325-024-03079-2. Epub 2024 Dec 23. PMID 39714546
- [Derived] Ogura T, Inoue Y, Azuma A, Homma S, Kondoh Y, Tanaka K, Ochiai K, Sugiyama Y, Nukiwa T. Real-World Safety and Tolerability of Nintedanib in Patients with Idiopathic Pulmonary Fibrosis: Interim Report of a Post-Marketing Surveillance in Japan. Adv Ther. 2023 Apr;40(4):1474-1493. doi: 10.1007/s12325-022-02411-y. Epub 2023 Jan 24. PMID 36692681
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-interventional study based on newly collected data aimed to evaluate safety and effectiveness of Ofev Capsules treatment in patients with Idiopathic Pulmonary Fibrosis (IPF) who newly initiated Ofev capsules under a real-world setting.
Pre-assignment Details: Only subjects that met all inclusion and none of the exclusion criteria were included.
  Patients diagnosed with idiopathic pulmonary fibrosis (IPF) based upon the most recent ATS/ERS/JRS/ALAT guideline and who initiated treatment with Ofev Capsules after the launch were registered into this study basically within 14 days from initiation of Ofev Capsules (from October 2015 to May 2023, following enrollment in August 31st).
Groups:
- IPF Patients Receiving Nintedanib: Patients diagnosed with idiopathic pulmonary fibrosis (IPF) based upon the most recent ATS/ERS/JRS/ALAT guideline and who initiated treatment with Ofev Capsules after the launch were registered into this study basically within 14 days from initiation of Ofev Capsules (from October 2015 to May 2023, following enrollment in August 31st).
Period: Overall Study
Arm/Group | IPF Patients Receiving Nintedanib
Started (registered patients) | 10117
Treated | 5753
Completed | 1535
Not Completed | 8582
Not completed — No data reliability | 1
Not completed — no patient visit | 18
Not completed — missing info in CRF | 13
Not completed — Withdrawal by Subject | 616
Not completed — Lost to Follow-up | 312
Not completed — Improved | 22
Not completed — Lack of Efficacy | 316
Not completed — Adverse Event | 2553
Not completed — Not treated | 1
Not completed — No CRF collected | 138
Not completed — without CRF | 4225
Not completed — Physician Decision | 367

BASELINE CHARACTERISTICS:
Population: Safety set: This patient set included all patients who didn't have any predefined important protocol deviations (IPDs) leading to exclusion from this analysis set.
Arm/Group | IPF Patients Receiving Nintedanib
Number analyzed (Participants) | 5734
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1256
  Male | 4478
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Any Suspected Adverse Drug Reactions (ADRs)
Description: Number of patients with any suspected Adverse Drug Reactions (ADRs) is presented.
Time Frame: Up to 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | IPF Patients Receiving Nintedanib
Number analyzed (Participants) | 5734
Participants | 3852

2. Secondary Outcome: Absolute Change From Baseline in Forced Vital Capacity (FVC) at Week 104
Description: Absolute change from baseline in Forced Vital Capacity (FVC) at Week 104 is presented.
  Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. It is measured in Milliliter by spirometry.
Time Frame: At baseline and at week 104
Population: Effectiveness set: This patient set included all patients with Ofev Capsules in the safety set who were suffering from the approved indication. Further important protocol deviations (IPDs) leading to exclusion from this analysis set were predefined. Only patients with FVC and %FVC value at baseline and post treatment in effectiveness set were included in this analysis.
Measure: Mean (Standard Deviation); unit: MilliLiter (mL)
Arm/Group | IPF Patients Receiving Nintedanib
Number analyzed (Participants) | 481
MilliLiter (mL) | -152.5 (323.0)

ADVERSE EVENTS:
Time Frame: Up to week 104
Description: Safety set: This patient set included all patients who didn't have any predefined important protocol deviations (IPDs) leading to exclusion from this analysis set.
Arm/Group | IPF Patients Receiving Nintedanib
All-Cause Mortality (participants affected / at risk) | 1137/5734
Serious Adverse Events (participants affected / at risk) | 2326/5734
Other Adverse Events (participants affected / at risk) | 3239/5734
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IPF Patients Receiving Nintedanib (N=5734)
Acquired haemophilia (Blood and lymphatic system disorders) | 1
Agranulocytosis (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 5
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 2
Myelosuppression (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Acute myocardial infarction (Cardiac disorders) | 6
Angina pectoris (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 2
Aortic valve stenosis (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 7
Atrial flutter (Cardiac disorders) | 1
Atrial thrombosis (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Atrioventricular block second degree (Cardiac disorders) | 1
Bundle branch block right (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac dysfunction (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 57
Cardiac failure acute (Cardiac disorders) | 4
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 15
Cardio-respiratory arrest (Cardiac disorders) | 18
Cardiogenic shock (Cardiac disorders) | 1
Cardiomegaly (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 1
Cor pulmonale (Cardiac disorders) | 5
Coronary artery stenosis (Cardiac disorders) | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 5
Myocardial ischaemia (Cardiac disorders) | 2
Pericarditis (Cardiac disorders) | 1
Prinzmetal angina (Cardiac disorders) | 2
Right ventricular dysfunction (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 12
Sinus node dysfunction (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia paroxysmal (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 2
Deafness (Ear and labyrinth disorders) | 2
Adrenal insufficiency (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 5
Cataract (Eye disorders) | 4
Epiretinal membrane (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Macular hole (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Tolosa-Hunt syndrome (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Anal fistula (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Colitis ischaemic (Gastrointestinal disorders) | 4
Colitis ulcerative (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Crohn's disease (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 52
Diverticular perforation (Gastrointestinal disorders) | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Duodenal perforation (Gastrointestinal disorders) | 4
Duodenal ulcer (Gastrointestinal disorders) | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 6
Food poisoning (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 10
Gastrointestinal mucosal exfoliation (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 4
Haematochezia (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Ileus paralytic (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 2
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal infarction (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 2
Large intestine perforation (Gastrointestinal disorders) | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Lower gastrointestinal perforation (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 6
Melaena (Gastrointestinal disorders) | 6
Mesenteric panniculitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Obstruction gastric (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 5
Peptic ulcer (Gastrointestinal disorders) | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1
Rectal ulcer (Gastrointestinal disorders) | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Volvulus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 2
Chest pain (General disorders) | 5
Chills (General disorders) | 1
Condition aggravated (General disorders) | 1
Death (General disorders) | 51
Decreased activity (General disorders) | 3
Disease progression (General disorders) | 1
General physical health deterioration (General disorders) | 11
Inflammation (General disorders) | 1
Malaise (General disorders) | 9
Multiple organ dysfunction syndrome (General disorders) | 4
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 18
Sudden cardiac death (General disorders) | 1
Sudden death (General disorders) | 6
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 4
Biliary colic (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 4
Cholangitis acute (Hepatobiliary disorders) | 3
Cholecystitis (Hepatobiliary disorders) | 13
Cholecystitis acute (Hepatobiliary disorders) | 5
Cholelithiasis (Hepatobiliary disorders) | 2
Drug-induced liver injury (Hepatobiliary disorders) | 23
Hepatic cirrhosis (Hepatobiliary disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 58
Jaundice (Hepatobiliary disorders) | 2
Liver disorder (Hepatobiliary disorders) | 38
Liver injury (Hepatobiliary disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Amyloidosis (Immune system disorders) | 1
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 9
Decreased immune responsiveness (Immune system disorders) | 1
Abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 3
Appendicitis perforated (Infections and infestations) | 1
Aspergilloma (Infections and infestations) | 1
Aspergillus infection (Infections and infestations) | 3
Atypical mycobacterial infection (Infections and infestations) | 3
Bacterial infection (Infections and infestations) | 2
Brain abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 18
Bronchitis bacterial (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 18
Cellulitis (Infections and infestations) | 3
Cholangitis infective (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Complicated appendicitis (Infections and infestations) | 1
Cryptococcosis (Infections and infestations) | 1
Diabetic gangrene (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 5
Enteritis infectious (Infections and infestations) | 2
Enterococcal infection (Infections and infestations) | 1
Enterocolitis bacterial (Infections and infestations) | 2
Fungal infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 5
Hepatitis B reactivation (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 8
Herpes zoster disseminated (Infections and infestations) | 1
Infection (Infections and infestations) | 7
Infectious pleural effusion (Infections and infestations) | 7
Influenza (Infections and infestations) | 22
Liver abscess (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 6
Meningitis cryptococcal (Infections and infestations) | 1
Mycobacterial infection (Infections and infestations) | 1
Mycobacterium avium complex infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 5
Oral fungal infection (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Pneumococcal infection (Infections and infestations) | 3
Pneumococcal sepsis (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 207
Pneumonia aspiration (Infections and infestations) | 58
Pneumonia bacterial (Infections and infestations) | 155
Pneumonia cytomegaloviral (Infections and infestations) | 1
Pneumonia fungal (Infections and infestations) | 2
Pneumonia influenzal (Infections and infestations) | 2
Pneumonia klebsiella (Infections and infestations) | 1
Pneumonia legionella (Infections and infestations) | 1
Pneumonia moraxella (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 8
Pneumonia staphylococcal (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 4
Pulmonary tuberculosis (Infections and infestations) | 3
Pyelonephritis (Infections and infestations) | 2
Pyelonephritis acute (Infections and infestations) | 1
Pyuria (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 25
Scedosporium infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 12
Septic shock (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Systemic candida (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 11
Viral infection (Infections and infestations) | 3
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 6
Femur fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Heat illness (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1
Open fracture (Injury, poisoning and procedural complications) | 1
Pancreatic leak (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Pneumoconiosis (Injury, poisoning and procedural complications) | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 4
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood pressure decreased (Investigations) | 3
Blood pressure increased (Investigations) | 1
Brain natriuretic peptide increased (Investigations) | 1
C-reactive protein increased (Investigations) | 9
Fibrin D dimer increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
Hepatic enzyme abnormal (Investigations) | 1
Hepatic enzyme increased (Investigations) | 6
KL-6 increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Liver function test increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 3
Oxygen saturation decreased (Investigations) | 3
Platelet count decreased (Investigations) | 13
Red blood cell morphology abnormal (Investigations) | 1
Weight decreased (Investigations) | 5
White blood cell count decreased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Cachexia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 67
Dehydration (Metabolism and nutrition disorders) | 11
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 9
Hypophagia (Metabolism and nutrition disorders) | 2
Marasmus (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Zinc deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1
Immobilisation syndrome (Musculoskeletal and connective tissue disorders) | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Periostitis (Musculoskeletal and connective tissue disorders) | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1
Polymyositis (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Sarcopenia (Musculoskeletal and connective tissue disorders) | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 2
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 55
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 82
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Altered state of consciousness (Nervous system disorders) | 5
Carotid artery occlusion (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 3
Cerebral infarction (Nervous system disorders) | 22
Cerebrovascular disorder (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 7
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 6
Encephalopathy (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 2
Facial paralysis (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2
Lacunar infarction (Nervous system disorders) | 2
Loss of consciousness (Nervous system disorders) | 4
Myelopathy (Nervous system disorders) | 1
Paralysis (Nervous system disorders) | 1
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Stupor (Nervous system disorders) | 5
Subarachnoid haemorrhage (Nervous system disorders) | 2
Thalamus haemorrhage (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 10
Depression (Psychiatric disorders) | 3
Eating disorder (Psychiatric disorders) | 2
Mania (Psychiatric disorders) | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Azotaemia (Renal and urinary disorders) | 1
Bladder perforation (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 2
Diabetic nephropathy (Renal and urinary disorders) | 2
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
IgA nephropathy (Renal and urinary disorders) | 2
Nephrotic syndrome (Renal and urinary disorders) | 5
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal disorder (Renal and urinary disorders) | 6
Renal failure (Renal and urinary disorders) | 4
Renal impairment (Renal and urinary disorders) | 7
Renal infarct (Renal and urinary disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 5
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 73
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 8
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 12
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 3
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1000
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 45
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 9
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 41
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 191
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 15
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 50
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 102
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4
Drug eruption (Skin and subcutaneous tissue disorders) | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 2
Lung transplant (Surgical and medical procedures) | 4
Prostatic operation (Surgical and medical procedures) | 1
Pulmonary resection (Surgical and medical procedures) | 1
Surgery (Surgical and medical procedures) | 1
Aortic aneurysm (Vascular disorders) | 1
Aortic dissection (Vascular disorders) | 1
Artery dissection (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 7
Embolism arterial (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Microscopic polyangiitis (Vascular disorders) | 2
Paradoxical embolism (Vascular disorders) | 1
Peripheral circulatory failure (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IPF Patients Receiving Nintedanib (N=5734)
Diarrhoea (Gastrointestinal disorders) | 2036
Nausea (Gastrointestinal disorders) | 347
Hepatic function abnormal (Hepatobiliary disorders) | 829
Liver disorder (Hepatobiliary disorders) | 437
Decreased appetite (Metabolism and nutrition disorders) | 579

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT02607722/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT02607722/SAP_001.pdf